CLINICAL TRIAL: NCT01244958
Title: Addition of Rituximab to Leflunomide in Patients With Active Rheumatoid Arthritis - a Multicenter Randomised Double-blind Clinical Trial
Brief Title: Addition of Rituximab to Leflunomide in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Frank Behrens (Other)
Responsible Party: Sponsor-Investigator, Frank Behrens, Dr. med Frank Behrens, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFM07-Rtx-Lef; 2009-015950-39 (EudraCT Number)
Record Dates: First submitted 2010-09-28; First posted 2010-11-22 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Active rheumatoid arthritis; leflunomide; rituximab; inadequate clinical response to leflunomide
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab 1000 mg (Active Comparator): Administration of 1000 mg Rituximab in Part I, followed by either re-treatment with 1000 mg Rituximab or with 500 mg Rituximab in Part II of the study
  Interventions: Biological: Rituximab
- Placebo (Placebo Comparator): Administration of Placebo in Part I followed by re-treatment with either 1000 mg Rituximab or with 500 mg Rituximab in Part II of the study
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Rituximab — 1000 mg Rituximab infusion
  Other Names: Mab Thera
  Arms: Rituximab 1000 mg
Drug: Placebo — infusion of Sodium citrate, Polysorbate, Sodium chloride
  Arms: Placebo

SUMMARY:
Combination of rituximab (RTX) with several different chemotherapeutic regimes has proven synergistic effects in patients with either lymphoma or autoimmune diseases. First data of uncontrolled trials with the combination of RTX and leflunomide (LEF) are available.

DETAILED DESCRIPTION:
Rituximab provides lasting improvement in the signs and symptoms of rheumatoid arthritis (RA) after two infusions per treatment course in tumor necrosis factor (TNF) inhibitor inadequate responder (IR) patients. Importantly, MabThera® has been shown to inhibit radiographic progression in this highly pre-treated patient population. Rituximab is licensed for adult patients with severe active RA in combination with methotrexate after inadequate response to previous treatment, including TNF alpha- Inhibitors.

In daily practice the combination with methotrexate is often limited to side effects or contraindications to Methotrexate (MTX). Therefore there is an unmet medical need for evidence for the combination of RTX with other Disease modifying anti-rheumatic drugs (DMARDs)than MTX.

Leflunomide is a DMARD that selectively inhibits de novo pyrimidine synthesis by blocking the enzyme dihydro-orotate dehydrogenase, thereby preventing DNA synthesis. The efficacy and safety of leflunomide in patients with active RA have been demonstrated in three phase III studies. Leflunomide was shown to be better than placebo and at least as effective as methotrexate in improving individual signs and symptoms of RA; these responses were seen as early as 4 weeks and were maintained for up to 2 years. Leflunomide was also effective in slowing disease progression as assessed by radiographic analysis of joint damage, and in improving functional activity as measured by the Stanford Health Assessment Questionnaire Disease Activity Index. An open label extension study of patients treated with leflunomide demonstrated that these improvements are maintained for up to 5 years in a subset of patients, with no new or unexpected adverse events emerging compared with the initial phase III studies.

In Europe leflunomide is often used in daily clinical practice as an alterative to MTX in patients with active RA.

Recently published data of a small open label trial (Vital et al. 2008) and data of a German non-interventional study (NIS) (Wendler et al. 2009) demonstrated the effectiveness of the addition of RTX to leflunomide in patients with active RA. The proportion of patients achieving EULAR (European League against Rheumatism) moderate to good response was 61% for RTX alone, 65 % for RTX plus MTX and 79% for RTX plus leflunomide in the German NIS. In the Leeds study of Vital et al.

33% of the patients achieved ACR (American College of Rheumatology)50 response (ACR 20: 68%, ACR 70: 20%) despite multiple pre-treatments, including patients with inadequate response to three TNF-Inhibitors.

The low rate of serious adverse drug reactions in the different groups of the German NIS demonstrated the safety of the combination of RTX and leflunomide (n=90) (1.6 / 1.1 / 0,5% for RTX+MTX / RTX+LEF / RTX Mono, 5.1 / 6,7 / 3,8% experienced infusion reactions)

ELIGIBILITY:
Inclusion Criteria:

Male and female patients, 18 to 75 years of age, with active rheumatoid arthritis (RA) who have had an inadequate response to disease modifying anti-rheumatic drugs, not more than 3 non-biological DMARDs including leflunomide, and not more than one inadequate response to anti-TNF-therapy, and currently have active disease despite at least 3-month treatment with leflunomide. Active disease is defined as DAS 28 >3.2 and at least swollen joint count (SJC) ≥ 3 and tender joint count (TJC) ≥ 3 included in the 28 joint count.

* Male and female patients with rheumatoid arthritis for at least 3 months diagnosed according to the revised 1987 ACR criteria for the classification of rheumatoid arthritis.
* Willingness and capability to give written informed consent, and willingness to participate and to comply with the study protocol.
* Not more than 2 non-biological DMARDs other than leflunomide in history, which are washed out at least 4 weeks prior to first rituximab infusion
* Previous use of anti-TNF therapy is allowed. Patient will only be allowed to be pre-treated with a maximum of two anti-TNF therapies and only one stopped due to inadequate response. The second anti-TNF could be stopped for instance due to intolerance, e.g. injection site reactions. Anti-TNF treatment must be discontinued prior to baseline considering the different characteristics of the specific compound: Use of infliximab, adalimumab, certolizumab, golimumab within 8 weeks of baseline, use of etanercept within 4 weeks of baseline.

Exclusion Criteria:

* RA functional class IV: limited in ability to perform usual self-care, work, and other activities
* Male and female patients with other chronic inflammatory articular disease or systemic autoimmune disease
* Any active infection, a history of recurrent clinically significant infection, a history of recurrent bacterial infections with encapsulated organisms (Hepatitis B, C and HIV (human immune deficiency virus) - will be tested at screening)
* Chronic, latent and acute infections of the lung
* Positive result of a Tuberculosis specific Interferon gamma release assay (will be tested at screening)
* Primary or secondary immunodeficiency
* History of cancer with curative treatment not longer than 5 years ago except basal-cell carcinoma of the skin that had been excised
* Evidence of significant uncontrolled concomitant diseases or serious and / or uncontrolled diseases that are likely to interfere with the evaluation of the patient's safety and of the study outcome
* Neuropathy that can interfere with filling out the patient's questionnaires
* History of a severe psychological illness or condition
* Known hypersensitivity to any component of the product or to murine proteins
* Severe heart failure (New York Heart Association Class III and IV) or severe,uncontrolled cardiac disease.
* Women lactating, pregnant, nursing or of childbearing potential with a positive pregnancy test or planned pregnancy.
* Women of childbearing potential without adequate contraception (medically acceptable methods (pearl Index < 1) are contraceptive implant, contraceptive injection, intrauterine device (IUD), or oral contraceptives taken for at least 3 months,which the patient agrees to continue using during the study, or a double-barrier method which must consist of a combination of any of the following: diaphragma,cervical cap, condom, or spermicide)
* History of alcohol, drug or chemical abuse (defined as impaired / questionable reliability) as well as neurotic personality.
* Participation in another investigational study within 4 weeks prior to the screening visit.
* Previous treatment with any B-cell depleting agents including rituximab
* Intolerance to ingredients of rituximab or murine proteins
* Pre-treatment with abatacept, tocilizumab or other anti-TNF biologicals.
* Inadequate response to more than one anti-TNF-therapy
* Pre-treatment of more than two anti-TNF, only one is allowed to be stopped due to inadequate response. The second anti-TNF could be stopped due to intolerance, e.g. injection site reactions
* Corticosteroids at doses exceeding 10 mg per day of prednisolone or equivalents within the last 2 weeks or corticosteroids at instable doses within the last 2 weeks
* Intolerance or contraindication to drugs required for the treatment of the side effects of rituximab
* Previous treatment with any investigational medicinal product within last 3 months prior to baseline
* Receipt of a live vaccine within 4 weeks prior to treatment
* Intra- articular or parenteral corticosteroids within 4 weeks prior to screening visit
* Haemoglobin < 8.5 g / dl (equivalent to < 5,28 mmol/l Haemoglobin)
* Neutrophil counts < 1.500 / μl (equivalent to 1,5 / nl)
* Platelet count < 75.000 / μl (equivalent to 75 / nl)
* Lower than 500 / μl (equivalent to 0,5 / nl) lymphocytes
* Serum creatinine > 1.4 mg / dl for women or 1.6 mg / dl for men
* Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) > 2.5 times upper limit of normal
* IgG (immunoglobulin G) level < 5g/l

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2010-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
ACR 50 - Part I of the Study - 50% improvement of ACR defined disease activity | Week 24
  Proportion of patients with an ACR 50 response at week 24
DAS28 - Part II of the study - evaluation of Disease activity score (DAS)28 | week 52
  Mean of DAS28 at week 52

SECONDARY OUTCOMES:
Evaluation of 50 % improvement of ACR defined disease activity (ACR 50) | From baseline (day of IMP administration) until up to 52 weeks
  To determine the efficacy and safety at week 24 of rituximab treatment of 2x1000 mg i.v. vs. placebo and the efficacy and safety at week 52 of rituximab 2x1000 mg i.v. vs 2x500 mg
EULAR response - response to therapy defined by European League against Rheumatism (EULAR) | From baseline (day of IMP administration) until up to 52 weeks
  EULAR response rates at week 16, 24, 40, 48
Assessment of ACR core set consisting of SJC, TJC, HAQ, patient's and physician's global assessments - Visual analog scales (VAS), Subject's pain-scale, CRP, ESR | From baseline (day of IMP administration) until up to 52 weeks
  Change in ACR core set (Swollen Joint count (SJC), Tender Joint Count (TJC), Health Assessment Questionnaire (HAQ), patient's and physician's global assessments visual analog Scale (VAS), subject's pain scale, C-reactive protein (CRP) and Erythrocyte sedimentation rate (ESR))compared to baseline at all follow-up visits
Assessment of SF-36 scores (Health survey) | From baseline (day of IMP administration) until up to 52 weeks
  Change in SF-36 scores compared to baseline at all followup visits
Assessment of FACIT (Functional assessment of chronical illness therapy)-fatigue- Questionnaire | From baseline (day of IMP administration) until up to 52 weeks
  Change in FACIT-fatigue assessment compared to baseline at all follow-up visits at week 16, 24, 40 and 48
HAQ (health assessment questionnaire)- assessment | From baseline (day of IMP administration) until up to 52 weeks
  Change in HAQ assessment compared to baseline at follow-up visits at week 8, 12, 16, 24, 32, (36), 40, 48, 52
proportion of DAS28-ESR remission - remission using DAS28 based on the erythrocyte sedimentation rate (ESR) defined as DAS28 < 2.6 | from week 16 until 48 weeks
  Proportion of patients achieving DAS28-ESR remission (DAS28 < 2.6) at week 16, 24, 40, 48
Proportion of patient with disease activity score in 28 joints (DAS28) based on the erythrocyte sedimentation rate (ESR) (DAS28-ESR) - low disease is defined DAS28 < 3.2 | from week 16 until 48 weeks
  Proportion of patients achieving DAS28-ESR low disease (DAS28 < 3.2) at week 16, 24, 40, 48
Assessment of changes in c-reactive protein (CRP) and Erythrocyte sedimentation rate (ESR) values | From baseline (day of IMP administration) until up to 52 weeks
  Change of CRP and ESR compared to baseline at all follow-up visits at week 2, 8, 12, 16, 24, 32, (36), 40, 48, 52
Assessment of changes in rheumatoid factor (RF) and Antibody against cyclic citrullinated peptide (aCCP) values | At Screening
  Change of RF and aCCP compared at Screening, 16, 24, and 48
Performance of standardized ultrasound synovitis score (US7)in subgroup of patients | From baseline (day of IMP administration) until up to 48 weeks
  Change in ultrasound synovitis score (if possible 3rd party blind observer, imaging subgroup only) performed at baseline and week 16, 24, 40, 48
Assessment of changes of rheumatoid nodules (number and diameter of target nodule) during therapy | From baseline (day of IMP administration) until up to 48 weeks
  Numbers of rheumatoid nodules and the diameter of one target nodule at baseline, week 24 and 48
Assessment of main safety parameters as SAE, deaths, duration of B-cell depletion and rate of infections + malignancies | From week 2 until up to 52 weeks
  Safety parameters:
  * Number of deaths, drop-out rates, causes of drop-outs, summary of SAEs per treatment group and severity of adverse events
  * Extent and duration of B cell depletion
  * Rates of infections, malignancies
Documentation of used standard care treatment by patients that are non-responder to therapy | Week 26
  Explorative analysis of the effect of standard care treatment in patients with insufficient response to the investigational medicinal product
Descriptive analysis of outcome measures in patients differentiated by presence of rheumatoid factor (RF-positive) or absence of rheumatoid factor(RF-negative) | At Screening
  Descriptive analysis of change in ACR20/50/70, EULAR Response and DAS28 in RF-positive and RF-negative patients, respectively
Assessment of changes in rheumatoid factor (RF) and Antibody against cyclic citrullinated peptide (aCCP) values | week 16
  Change of RF and aCCP compared at Screening, 16, 24, and 48
Assessment of changes in rheumatoid factor (RF) and Antibody against cyclic citrullinated peptide (aCCP) values | week 24
  Change of RF and aCCP compared at Screening, 16, 24, and 48
Assessment of changes in rheumatoid factor (RF) and Antibody against cyclic citrullinated peptide (aCCP) values | week 48
  Change of RF and aCCP compared at Screening, 16, 24, and 48
Assessment of changes of rheumatoid nodules (number and diameter of target nodule) during therapy | week 24
  Numbers of rheumatoid nodules and the diameter of one target nodule at baseline, week 24 and 48
Assessment of changes of rheumatoid nodules (number and diameter of target nodule) during therapy | week 48
  Numbers of rheumatoid nodules and the diameter of one target nodule at baseline, week 24 and 48
Documentation of used standard care treatment by patients that are non-responder to therapy | Week 36
  Explorative analysis of the effect of standard care treatment in patients with insufficient response to the investigational medicinal product
Documentation of used standard care treatment by patients that are non-responder to therapy | Week 48
  Explorative analysis of the effect of standard care treatment in patients with insufficient response to the investigational medicinal product
Descriptive analysis of outcome measures in patients differentiated by presence of rheumatoid factor (RF-positive) or absence of rheumatoid factor(RF-negative) | week 16
  Descriptive analysis of change in ACR20/50/70, EULAR Response and DAS28 in RF-positive and RF-negative patients, respectively
Descriptive analysis of outcome measures in patients differentiated by presence of rheumatoid factor (RF-positive) or absence of rheumatoid factor(RF-negative) | week 24
  Descriptive analysis of change in ACR20/50/70, EULAR Response and DAS28 in RF-positive and RF-negative patients, respectively
Descriptive analysis of outcome measures in patients differentiated by presence of rheumatoid factor (RF-positive) or absence of rheumatoid factor(RF-negative) | week 48
  Descriptive analysis of change in ACR20/50/70, EULAR Response and DAS28 in RF-positive and RF-negative patients, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Frank Behrens, Dr. med., Principal Investigator — Department of Medicine II / Rheumatology Johann Wolfgang Goethe-Universität
Locations (45):
- Germany (45):
  - Schwerpunktpraxis, Bad Kösen, Saxony-Anhalt
  - Kerckhoff-Klinik GmbH Abtlg. Rheumatologie und Klin. Immunologie, Bad Nauheim
  - Rheumazentrum Baden-Baden, Baden-Baden
  - Praxis Remstedt, Berlin
  - Rheumaklinik Berlin-Buch Immanuel Krankenhaus, Berlin
  - Schlosspark-Klinik, Berlin
  - Universitätsmedizin Berlin-Campus Charité, Berlin
  - Krankenhaus Porz am Rhein, Cologne
  - Universitätsklinikum Köln Med I, Cologne
  - Krankenhaus Friedrichstadt, Dresden
  - Rheumatologische Schwerpunktpraxis, Erlangen
  - Department of Medicine II / Rheumatology Johann Wolfgang Goethe-Universität, Frankfurt
  - Rheumatologie Endokrinologikum Frankfurt, Frankfurt
  - Universität Freiburg Innere Medizin - Abtlg. Rheumatologie, Freiburg im Breisgau
  - Gemeinschaftspraxis für Innere Medizin, Giessen
  - Praxis, Innere Medizin und Rheumatologie, Goslar
  - Universitätsmedizin Göttingen Georg-August-Universität Abtlg. Nephrologie u. Rheumatologie, Göttingen
  - Klinik u. Poliklinik f. Innere Medizin A, Nephrologie u. Rheumatolog Uniklinik Greifswald, Greifswald
  - Uniklinik Halle - Poliklinik für Innere Medizin I, Halle
  - Medizinische Hochschule Hannover Klinik f. Immunologie u. Rheumatologie, Hanover
  - Rheumapraxis Heidelberg, Heidelberg
  - Praxis, Innere Medizin und Rheumatologie, Hildesheim
  - Internistisch - Rheumatologische Praxis, Hofheim
  - Klinik für Innere Medizin I Universitätsklinikum des Saarlandes, Homburg
  - Rheumapraxis Karlsruhe, Karlsruhe
  - Universität Leipzig, Leipzig
  - Praxis Kaufmann, Ludwigsfelde
  - Medizinsche Klinik A, Rheumatologie, Nephrologie Klinikum der Stadt Ludwigshafen,, Ludwigshafen
  - Katholisches Klinikum Mainz, St. Vincenz und Elisabeth Hospital, Mainz
  - Praxis Prof. Dr. Kellner, München
  - Praxiszentrum St. Bonifatius, München
  - Rheumatologische Schwerpunktpraxis, Neuss
  - Klinikum Offenbach GmbH, Offenbach
  - Praxis. Gauler und Fliedner, Osnabrück
  - Praxis Gräßler, Pirna
  - Rheumatologie Praxis, Planegg
  - Evangelisches Fachkrankenhaus, Ratingen
  - Uni Klinik Regensburg, Regensburg
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Abt. II Medizinische Universitätsklinik und Poliklinik, Tübingen
  - Universitätsklinikum Ulm Klinik f. Innere Medizin III, Ulm
  - Innere Medizin und Rheumatologie, Villingen-Schwenningen
  - Rheumatologische Praxis Dr. Wörth, Wiesbaden
  - Rheumatologische Schwerpunktpraxis, Wuppertal
  - Med. Klinik und Poliklinik III, Schwerpunkt Rheumatologie, Würzburg

REFERENCES:
- [Derived] Koehm M, Foldenauer AC, Rossmanith T, Alten R, Aringer M, Backhaus M, Burmester GR, Feist E, Kellner H, Krueger K, Muller-Ladner U, Rubbert-Roth A, Tony HP, Wassenberg S, Burkhardt H, Behrens F. Effectiveness of Different Rituximab Doses Combined with Leflunomide in the Treatment or Retreatment of Rheumatoid Arthritis: Part 2 of a Randomized, Placebo-Controlled, Investigator-Initiated Clinical Trial (AMARA). J Clin Med. 2022 Dec 9;11(24):7316. doi: 10.3390/jcm11247316. PMID 36555933
- [Derived] Behrens F, Koehm M, Rossmanith T, Alten R, Aringer M, Backhaus M, Burmester GR, Feist E, Herrmann E, Kellner H, Krueger K, Lehn A, Muller-Ladner U, Rubbert-Roth A, Tony HP, Wassenberg S, Burkhardt H. Rituximab plus leflunomide in rheumatoid arthritis: a randomized, placebo-controlled, investigator-initiated clinical trial (AMARA study). Rheumatology (Oxford). 2021 Nov 3;60(11):5318-5328. doi: 10.1093/rheumatology/keab153. PMID 33738492